CLINICAL TRIAL: NCT03892330
Title: A Multicenter, Randomized, Double-blind, Prospective Study to Evaluate the Efficacy and Safety of Vincristine, Dactinomycin/Cyclophosphamide Combination Therapy Combined With Liposomal Doxorubicin/Doxorubicin/Pharmorubicin/Pirarubicin in 0.5-14 Year Old Children With Nephroblastoma.
Brief Title: Combination Therapy of Anthracyclines for Children With Nephroblastoma
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Weisong Cai, Professor, Shengjing Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SJZE001
Record Dates: First submitted 2019-03-25; First posted 2019-03-27 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: 0.5-14 Year Old Children With Nephroblastoma
Keywords: Nephroblastoma; Anthracycline; Liposome doxorubicin; Doxorubicin; Pharmorubicin; Pirarubicin
MeSH Terms: conditions — Wilms Tumor | interventions — Vincristine; Oxytetracycline; Cyclophosphamide; liposomal doxorubicin; Doxorubicin; Epirubicin; pirarubicin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- liposomal doxorubicin (Experimental): Drugs: liposome doxorubicin Combination therapy: vincristine and dactinomycin or cyclophosphamide
  Interventions: Drug: Vincristine; Drug: Oxytetracycline/ Cyclophosphamide; Drug: Liposomal doxorubicin
- doxorubicin (Active Comparator): Drug: doxorubicin Combination therapy: vincristine and dactinomycin or cyclophosphamide
  Interventions: Drug: Vincristine; Drug: Oxytetracycline/ Cyclophosphamide; Drug: Doxorubicin
- pharmorubicin (Active Comparator): Drug: pharmorubicin Combination therapy: vincristine and dactinomycin or cyclophosphamide
  Interventions: Drug: Vincristine; Drug: Oxytetracycline/ Cyclophosphamide; Drug: Pharmorubicin
- pirarubicin (Active Comparator): Drug: pirarubicin Combination therapy: vincristine and dactinomycin or cyclophosphamide
  Interventions: Drug: Vincristine; Drug: Oxytetracycline/ Cyclophosphamide; Drug: Pirarubicin

INTERVENTIONS:
Drug: Vincristine — Dosage according to Children Wilms tumor diagnosis and therapy recommendations: Wilms Tumor-2016 (WT-2016) (2-6) Chemotherapy.
Drug: Oxytetracycline/ Cyclophosphamide — Dosage according to Children Wilms tumor diagnosis and therapy recommendations: Wilms Tumor-2016 (WT-2016) (2-6) Chemotherapy.
Drug: Liposomal doxorubicin — The dosage of Liposomal doxorubicin is half of doxorubicin dosage in Children Wilms tumor diagnosis and therapy recommendations: Wilms Tumor-2016 (WT-2016) (2-6) Chemotherapy.
  Arms: liposomal doxorubicin
Drug: Doxorubicin — Dosage according to Children Wilms tumor diagnosis and therapy recommendations: Wilms Tumor-2016 (WT-2016) (2-6) Chemotherapy.
  Arms: doxorubicin
Drug: Pharmorubicin — The dosage of pharmorubicin is 2 times of doxorubicin dosage in Children Wilms tumor diagnosis and therapy recommendations: Wilms Tumor-2016 (WT-2016) (2-6) Chemotherapy.
  Arms: pharmorubicin
Drug: Pirarubicin — The dosage of pirarubicin is equal to doxorubicin dosage in Children Wilms tumor diagnosis and therapy recommendations: Wilms Tumor-2016 (WT-2016) (2-6) Chemotherapy.
  Arms: pirarubicin

SUMMARY:
This study aims to estimate the efficacy and side effects of study drugs in children with nephroblastoma who are treated with combination therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age 6 months old to 14 years old.
2. No smoking history.
3. Pathologically confirmed nephroblastoma.
4. Informed consent and assent has been obtained before any study assessment is performed.
5. Good compliance.
6. Need to be applied to anthracycline chemotherapy according to the diagnosis and treatment recommendations for Chinese children with nephroblastoma (current version CCCG-WT-2016).
7. Need to be applied to doxorubicin according to the diagnosis and treatment recommendations for children with nephroblastoma (CCCG-WT-2016).

Exclusion Criteria:

1. Patients with cardiovascular disease in addition to nephroblastoma.
2. Patients with digestive, neurological, circulatory, renal or liver disease, blood disorders or growth abnormalities unrelated to the tumor.
3. Patients have been treated with chemotherapy or cardiotoxic nephrotoxic drugs in the past 4 weeks.
4. Patients have participated in other clinical trials in the past 4 weeks.
5. Patients with mediastinal disease.
6. Patients who have undergone mediastinal radiotherapy due to other tumors or received other treatments that may cause heart damage.

Ages: 6 Months to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2045-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 5 years
Time to treatment failure (TTF) | 5 years
Five-year Event free survival (5-year EFS) | 5 years

SECONDARY OUTCOMES:
Overall survival (OS) | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Shenjing Hospital, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided
Dear Sir/Madam Our study receives a grant from China Ministry of Science and Technology. We cannot decide whether the data could be shared. Hope you can understand.